CLINICAL TRIAL: NCT01399034
Title: Host DNA Methylation Patterns in Association With Periodontal Disease : MiRNA Changes in Obesity
Brief Title: Epigenetics, DNA Methylation Patterns and Periodontal Disease
Acronym: SZU
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Steven Offenbacher, DDS, MS, PhD, Center for Oral and Systemic Diseases
Other Study IDs: 07-0749; 1R01DE021052-01 (NIH)
Record Dates: First submitted 2011-07-12; First posted 2011-07-21 (Estimated); Last update posted 2011-07-21 (Estimated); Status verified 2011-07

CONDITIONS: Periodontal Disease
Keywords: Epigenomics; DNA methylation; MicroRNA; Periodontitis; Inflammation; Obesity
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Inflammation; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — * Gingiva biopsy samples (epithelium, connective tissue)
  * Gingival crevicular fluid
  * Saliva
  * Plaque samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- MicroRNA study: Obese group (+ periodontitis group) Non-obese group (+ periodontitis group)
- DNA methylation study: Periodontitis group Healthy periodontium group

SUMMARY:
The overall goal of this research is (1) to identify changes in gene expression and DNA methylation status in subjects who exhibit advanced chronic periodontal inflammation and (2) to identify microRNAs (miRNAs) and the interactive pathways associated with obesity as a modifier of periodontal infection pathogenesis.

DETAILED DESCRIPTION:
Aim 1. To determine whether diseased periodontal tissues biopsied from patients with periodontal disease will have altered DNA methylation patterns of selected genes as compared to the DNA methylation status biopsies obtained from adjacent, non-diseased periodontal sites, as well as periodontal biopsy samples obtained from non-diseased, healthy subjects.

Aim 2. To determine the role of tissue DNA Methylation on mRNA expression:

* 2a. To determine whether alterations in tissue mRNA expression (as determined by quantitative PCR) are associated with an aberrant DNA methylation status of respective gene promoter CpG islands in tissue biopsy samples obtained from diseased and non-diseased tissues from patients with periodontal disease and from non-diseased healthy subjects.
* 2b. By performing laser capture microdissection of biopsy samples from diseased patients [(epithelium, connective tissue and inflammatory infiltrate)] we seek to determine cellular patterns of mRNA expression and DNA methylation of targeted genes comparing inflamed to non-inflamed sites within diseased patients.
* 2c. We will perform in vitro studies to analyze whether gingival fibroblasts from patients with periodontal disease will show a differential methylation pattern and whether these cells will display a differential inflammatory response when compared to control fibroblasts isolated from healthy subjects.

Aim 3. The aim of this pilot investigation was to determine if miRNA expression differed in the presence or absence of obesity, comparing gingival biopsies obtained from patients with or without periodontal disease.

* 3a. To determine whether diseased periodontal tissues biopsied from patients with periodontal disease will influence the level of miRNA expression as compared to the biopsies obtained from non-diseased, healthy subjects.
* 3b. To determine whether BMI [nonobese subjects BMI <30kg/m2, obese subjects >30kg/m2] will influence the level of miRNA expression in biopsies from diseased periodontal tissues as compared to periodontal biopsy samples obtained from non-diseased, healthy subjects.

Gingival samples, gingival crevicular fluid, saliva and plaque samples will be collected and a periodontal examination will be performed. The periodontal assessment will record pocket depth, clinical attachment level and percent bleeding on probing. Blood pressure, height and weight (Body Mass Index assessment) will be obtained on participants as well.

Tissue gene expression by quantitative PCR and DNA methylation sequence analysis, proteomic analyses of gingival crevicular fluid, Differential Methylation Hybridization and, microRNA expression profile by Human miRNA Microarray and Real-time PCR quantification will all be performed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be adult males or females between the ages of 18 and 65 years (inclusive).
* Subjects must be able and willing to follow study procedures and instructions.
* Subjects must have read, understood and signed an informed consent form.
* Subjects must present with at least 20 teeth in the functional dentition, excluding third molars.
* Subjects must be in good general health.
* Subjects must present with advanced chronic periodontitis (American Dental Association Class 4) as determined by the investigator or designee during the screening periodontal examination. Such subjects will exhibit periodontal pocketing (>5 mm and Bleeding on Probing) and severe alveolar bone loss. Subjects will be under active care for periodontitis and will be treatment planned for periodontal flap surgery.
* Control subjects must present with periodontal health as determined by the investigator or designee during the screening periodontal examination. Such subjects will exhibit no evidence of periodontal pocketing (pockets ≤4mm), and no bleeding on probing at the site of the biopsy. Patients from this group will be treatment planned for routine crown extension procedures for restorative reasons, or be volunteers from the general population meeting the inclusion criteria.
* 24 subjects from group 2 will be enrolled based on Body Mass Index (BMI). Twelve obese subjects (BMI of 30 or greater) and twelve non-obese subjects (BMI less than 30) will be enrolled. Twelve from the obese and twelve from the non-obese group will be split in half based on periodontal status.
* 6 periodontal healthy non-obese
* 6 periodontal healthy obese
* 6 periodontal diseased non-obese
* 6 periodontal diseased obese

Exclusion Criteria:

* Individuals who have a chronic disease with oral manifestations.
* Individuals who exhibit gross oral pathology.
* Treatment with antibiotics for any medical or dental condition within 1 month prior to the screening examination.
* Chronic treatment (i.e., two weeks or more) with any medication known to affect periodontal status (e.g., phenytoin, calcium antagonists, cyclosporin, coumadin, non-steroidal anti-inflammatory drugs, aspirin) within one month of the screening examination.
* Ongoing medications initiated less than three months prior to enrollment (i.e., medications for chronic medical conditions must be initiated at least three months prior to enrollment).
* Subjects with clinically significant organ disease including impaired renal function, or any bleeding disorder.
* Subjects with active infectious diseases such as hepatitis, HIV or tuberculosis.
* Severe unrestored caries, or any condition that is likely to require antibiotic treatment over the trial, including the need for prophylactic antibiotic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ninety-eight subjects will be recruited from the Graduate Periodontics Clinic and Dental Faculty Practice at the University of North Carolina School of Dentistry and if needed from the general population. Subjects must present with either chronic periodontitis or periodontal health.
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2007-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
DNA methylation patterns of selected candidate genes | Visit 1

SECONDARY OUTCOMES:
Identification of miRNA species | Visit 1

CONTACTS AND LOCATIONS:
Overall Officials: Steven Offenbacher, DDS, MS, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Center for Oral and Systemic Diseases, Chapel Hill, North Carolina, United States